CLINICAL TRIAL: NCT05071547
Title: Internet-Delivered Acceptance And Commitment Therapy Added To Multimodal Pain Rehabilitation: A Cluster Randomized Controlled Pilot And Feasibility Trial
Brief Title: Guided Internet-delivered Psychological Treatment for Chronic Pain
Acronym: MERIT
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Linkoeping University (Other Government)
Responsible Party: Principal Investigator, Nina Bendelin, Principal investigator, PhD candidate, Lic. psychologist, Lic. psychotherapist, Msc., Linkoeping University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2010/186-31
Record Dates: First submitted 2021-09-10; First posted 2021-10-08 (Actual); Last update posted 2021-10-08 (Actual); Status verified 2021-09

CONDITIONS: Chronic Pain
Keywords: Internet-delivered Acceptance and Commitment Therapy (IACT); Interdisciplinary pain Rehabilitation Program (IRPR); Aftercare; Combined treatment
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Intervention Model Description: Upon acceptance and after informed consent has been obtained, participants are consecutively randomized to one of two study groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Internet-delivered acceptance and commitment therapy addition (Experimental): The IACT addition supplies participants with weekly educational material and additional exercises in line with live IRPR, although enriched with multimedia. Participants will have access to their rehabilitation content via the web-site and can practice in their homes in-between live sessions of IRPR.
  Interventions: Behavioral: Guided internet-delivered acceptance and commitment therapy (ACT)
- Interdisciplinary pain rehabilitation program (Active Comparator): A 6-week long multimodal treatment including approximately 108 hours on site, focusing on return to work. Psychologists, physicians, physiotherapists (PT) and occupational therapists (OT) give synchronized treatments with a CBT/ACT approach.
  Interventions: Other: Interdisciplinary Pain Rehabilitation Program (IPRP)

INTERVENTIONS:
Behavioral: Guided internet-delivered acceptance and commitment therapy (ACT) — ACT builds on cognitive behavioral therapy (CBT), and includes methods for experiential learning and focus on psychological flexibility
  Arms: Internet-delivered acceptance and commitment therapy addition
Other: Interdisciplinary Pain Rehabilitation Program (IPRP) — Multimodal treatment where physio therapists, occupational therapists, psychologists and physicians give synchronized treatments to raise physical and psychological function and promote return to work
  Arms: Interdisciplinary pain rehabilitation program

SUMMARY:
The aim of this feasibility study is to investigate if an addition of an internet-delivered psychological treatment, Acceptance and commitment therapy (IACT), can enhance the effect of an existing evidence-based interdisciplinary rehabilitation program (IRPR) for chronic pain patients enrolled in clinical tertiary care, on pain-related psychological outcomes. The study might contribute to developing internet-delivered treatments suitable for this patient group and also help develop implementation strategies for internet interventions in clinical services. The study is planned to run for 2 years and include 300 patients, of which 150 will be in the intervention group and 150 in the control condition.

The overall hypothesis is that the IACT addition will lead to better and more sustained results compared to the IRPR alone. The first sub-hypothesis is that the IACT addition will enhance adherence and uptake during the IRPR. The second sub-hypothesis is that the IACT addition will help patients maintain results after the IRPR has ended.

DETAILED DESCRIPTION:
The trial is an un-blinded single-center randomized controlled trial with two parallel study groups set at a clinical service in regular care at a University Hospital. An online true random-number service (www.random.org) executed by a research assistant not otherwise involved in the trial, will allocate participants, with 1:1 allocation ratio, upon enrollment. Patients will be recruited from a specialist pain clinic which provides tertiary care (IPRP) for non-malign chronic pain with mild to moderate psychiatric comorbidities and serves as competence center for complex chronic pain in its City Council in southern Sweden. As an active comparator will be used as the control condition, an effect size of d=0.30 (specific component comparator was expected. Given 80 % power and a 5% significance level, the sample size calculation indicated that 90 participants in each group were needed. Considering a 50% dropout rate, a sample size of 135 participants in each group would be sufficient. The study planned to include n=300. Outcome variables will be collected digitally on 4 occasions; at pre and post treatment, at post aftercare intervention and at 1 year follow up. Additional complementary pen-and-paper data will be drawn from a national register (the SQRP) at three occasions; at pre-baseline/enrollment, at post treatment and at 1 year follow up. Outcome measures include psychological outcomes: pain acceptance, psychological inflexibility, self-efficacy, harm/negative effects and psychosocial consequences of living with pain. Also, measures of cost-effectiveness, usability, dose and time spent will be collected. Patients with long pain duration, high pain intensity, overuse of analgesics, alcohol or opioids, social withdrawnness, depression, or previous treatment failures constitute high risk of attrition. Early signs of attrition will be monitored by delayed response frequency. A plan to prevent attrition will be set at the inclusion assessment. As long as participant follow the IPRP through, data will likely be collected and there will be opportunities to discuss or prevent drop-out. Data will be entered and stored digitally. The process is monitored by a responsible research assistant who will also alert the research time of missing data. Access to study data will be restricted to the research team.The two study arms will be compared using parametric methods for data analysis or other methods depending on the robustness of the data. Missing data will be handled depending on the robustness of the data, assessed by Little MCAR test. Intention to treat analysis is an opportunity given the missing is not more than 40 %. Mixed models may be an option given missing data is not random. The steering committee will act as data monitoring committee (the lead investigator excluded) and will decide of interim analyses and execute stopping guidelines. The research assistant responsible for data management will alert the steering committee if collected data on negative experiences of treatment signals that any participant needs additional care related to experiences of the trial. Any modifications to the protocol which may impact on the study, will be agreed on within the research group. These changes will be either documented to be addressed at publication or communicated with the regional Ethical board if needed. Written informed consent will be obtained as pre-measurement are collected. An oral consent will be obtained prior to that, during the assessment interview, whereas participants may ask for further information. All recruited participants will be given an identification number. As little personal information as possible (e.g. only informed consent forms) will be kept locally as the majority of participants' information will be digital, secured with password-protected access systems. The research team members will be given access to the cleaned data set. To ensure confidentiality, data dispersed to project team members will be blinded of any identifying participant information. The steering committee will have access to the un-cleaned data set. Post-trial care will be given by IPRP staff when needed.

ELIGIBILITY:
Inclusion criteria:

1. chronic pain (ie consistent for 6 months), w/out common comorbid or multimorbid diagnoses
2. awaiting start of IPRP after medical and psychiatric assessment
3. completion of informed consent and pre-measurement forms

Exclusion criteria:

1. unable to communicate in writing in Swedish
2. lack access to a smart phone, tablet or computer

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2010-11-01 (Actual); Primary Completion 2014-05-01 (Actual); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in pain acceptance (The Chronic Pain Acceptance Questionnaire, CPAQ) | Week 0 (pre treatment), week 6 (post treatment), week 17 (post aftercare) and at 1 year follow up.
  CPAQ is a measure of pain acceptance with 20 items rated on a 6-point scale ranging from "never true" to "always true" and divided into two subscales: activity engagement and pain willingness. CPAQ has been validated for a Swedish sample and for an internet sample. Studies have shown high test-retest reliability (α=0.72-0.92).

SECONDARY OUTCOMES:
Change in psychological inflexibility (Psychological Inflexibility in Pain Scale, PIPS) | Week 0 (pre treatment), week 6 (post treatment), week 17 (post aftercare) and at 1 year follow up.
  Twelve items are rated on a 7-point scale ranging from "never true" to "always true" and divided into two subscales: Avoidance and Cognitive fusion. Higher score means higher psychological inflexibility. PIPS has been found a valid and reliable measure which may function as a working mechanism in ACT for chronic pain

CONTACTS AND LOCATIONS:
Overall Officials: Björn Gerdle, PhD, Study Director — Pain and Rehabilitation Centre, and Department of Health, Medicine and Caring Sciences, Linköping University, Sweden

IPD SHARING:
Plan to Share IPD: No